CLINICAL TRIAL: NCT01772979
Title: Phase II Study With Trabectedin (Yondelis®) in BRCA1 and BRCA2 Mutation Carrier and BRCAness Phenotype Advanced Ovarian Cancer Patients
Brief Title: Study With Trabectedin in BRCA1 and BRCA2 Mutation Carrier and BRCAness Phenotype Ovarian Cancer
Acronym: MITO15
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Professor Giovanni Scambia, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MITO15
Record Dates: First submitted 2012-11-17; First posted 2013-01-21 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2012-12

CONDITIONS: BRCA1 and BRCA2 Mutation Carrier and BRCAness Phenotype
Keywords: Trabectedin; BRCA1 and BRCA2; BRCAness; Ovarian cancer
MeSH Terms: conditions — Fanconi Anemia, Complementation Group D1; Ovarian Neoplasms | interventions — Trabectedin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trabectedin (Experimental): Trabectedin 1.3 mg/m2 q 21 days
  Patients will receive trabectedin until disease progression or unacceptable toxicity
  Interventions: Drug: Trabectedin

INTERVENTIONS:
Drug: Trabectedin
  Other Names: Yondelis

SUMMARY:
This is a multicenter phase II study on trabectedin in advanced or recurrent ovarian cancer patients with BRCA mutation and BRCAness phenotype.

The purpose of this study is to determine the feasibility in terms of objective response rate by RECIST version 1.1 (Complete and Partial Response [CR + PR]) with trabectedin in patients with BRCA1 or BRCA2 mutation carrier or BRCAness phenotype advanced ovarian cancer patients.

DETAILED DESCRIPTION:
The main contribution to hereditary ovarian cancer comes from breast cancer (BRCA) genes mutations, which are responsible of 90% of hereditary ovarian cancer. The two susceptibility genes associated with epithelial-type OC are BRCA1 and BRCA2.

The BRCA proteins play an important role in the DNA repair mechanisms and are also involved in the control of the cell cycle checkpoints, in protein ubiquitinization and chromatin remodelling.

Mutations in the BRCA genes have been extensively described in families affected by breast and/or OC; mutated BRCA1 has been found in up to 75% of families with hereditary OC - Recent data suggest that dysfunction of BRCA1andBRCA2, so-called BRCAness, maybe more prevalent than originally assumed. Both genetic and epigenetic mechanisms can create the BRCAness phenotype in at least a third of all epithelial ovarian cancers. The definition of BRCAness ovarian cancer is: high-grade serous cancers, high initial sensitivity to platinum drugs and retention of platinum-sensitivity through multiple relapses, longer history of disease, longer survival, longer TFIs between relapses.

Yondelis® (trabectedin) is proposed to block the transcriptional activation of a subset of inducible genes without affecting their constitutive expression. Trabectedin binds to the minor groove of DNA, bending the helix to the major groove. This binding to DNA triggers a cascade of events affecting several transcription factors, DNA binding proteins, and DNA repair pathways, resulting in perturbation of the cell cycle.

Cell cycle studies of the action of trabectedin on tumor cells in vitro reveal that it decreases the rate of progression of the cells through S phase towards G2 and causes a prolonged blockade in G2/M at biologically relevant concentrations (20-80 nM). These cell cycle blocks are p53-independent and lead to a strong apoptopic response. Cells in G1 are more sensitive to the cytotoxic effects of trabectedin. These effects appear to be related to the unique 3-subunit structure, where two of the subunits or rings are involved in binding to the minor groove of DNA in guanine-cytosine rich sequences and alkylation N2 of guanine forming adducts that distorted the DNA helix structure and they are recognized by the TC-NER mechanism.

DNA repair proficiency is a major determinant for the cytotoxicity of trabectedin: human cell lines deficient for genes essential for TC-NER activity as XPA, XPB, XPD, XPF, XPG, ERCC1, CSA and CSB are resistant to trabectedin, and this resistance is reverted by complementation of the cells with the corresponding gene. Trabectedin induces double strand breaks and that the BRCA1-/- human cell line HCC1937 and BRCA2Δ22/Δ22 mice cells are more sensitive to trabectedin and this hypersensitivity is reverted by complementation by the BRCA1 or BRCA2 gene.

Based in these observations it was hypothesized that the NER machinery trapped in the DNA lesion induced by trabectedin was resolved by the cells producing double strand breaks that were repaired by the HRR machinery, and synergistic action of TC-NER and HRR machinery would be necessary for maximal trabectedin cytotoxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with partially platinum sensitive ovarian cancer (platinum-free interval 6-12 months) who have previously received at least two platinum based chemotherapy lines, BRCA mutated or with BRCAness phenotype.

   * Definition of BRCAness phenotype: high-grade serous cancers, great initial sensitivity to platinum drugs and retention of platinum-sensitivity through multiple relapses, long history of disease, long survival, long TFIs between relapses (patients with high personal risk factors will be included after doing the analysis for BRCA 1-2 mutation before knowing the results).
   * BRCA 1 and/or BRCA 2 mutation carriers (patients with established mutation will be included, patients with high personal risk factors will be included after doing the analysis before knowing the results)
2. Patients with platinum resistant ovarian cancer, BRCA mutated or with BRCAness phenotype who have previously received at least two previous chemotherapy lines (including platinum rechallenge).

   Definition of platinum resistant: Tumor progression within 6 months of completion of platinum-based therapy (after platinum re-challenge for platinum sensitive recurrence).
3. Patient's written informed consent before any clinical trial-specific procedure.
4. 18 years-of-age or older.
5. Measurable disease as defined in the Response Evaluation Criteria in Solid Tumors (RECIST) Guidelines
6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1.
7. Hematologic variables:

   1. Hemoglobin ≥9 g/dL
   2. Absolute neutrophil count (ANC) ≥1,500/μL, and
   3. Platelet count ≥100,000/μL.
8. Serum creatinine ≤ 1.5 mg/dL or creatinine clearance ≥ 30 mL/min
9. Creatinine phosphokinase (CPK) ≤ 2.5 ULN.
10. Hepatic function variables

    1. Total bilirubin ≤ ULN.
    2. Total alkaline phosphatase ≤ 2.5 ULN
    3. AST (serum aspartate transaminase [SGOT]) and ALT (serum alanine transaminase [SGPT]) must be ≤2.5 x ULN.
11. Albumin ≥ 25 g/l.
12. Adequately recovered from the acute toxicity of any prior treatment. -

Exclusion Criteria:

* 1. Prior exposure to trabectedin. 2. Known hypersensitivity to any of the components of the trabectedin i.v. formulation or dexamethasone.

  3. Less than 2 prior chemotherapy lines given in patients with partially platinum sensitive, BRCA mutated or BRCAness phenotype, ovarian cancer recurrences (including platinum rechallenge).

  4. Patients with platinum refractory, BRCA mutated or with BRCAness phenotype, ovarian cancer.

  5. Less than 4 weeks from last dose of therapy with any investigational agent, or chemotherapy.

  6. History of another neoplastic disease (except basal cell carcinoma or cervical carcinoma in situ adequately treated) unless in remission for 3 years or longer.

  7. Known clinically relevant CNS metastases. 8. Other serious illnesses, such as:

  • Congestive heart failure or angina pectoris; myocardial infarction within 1 year before enrollment; uncontrolled arterial hypertension or arrhythmias
  * Psychiatric disorder that prevents compliance with protocol
  * Active viral hepatitis; or chronic liver disease
  * Active infection
  * Any other unstable medical conditions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
objective response | 24 months
  To evaluate the feasibility (in terms of objective response rate by RECIST version 1.1) of Yondelis treatment in recurrent ovarian cancer population selected for BRCA mutation or BRCAness phenotype.
  The response rate will be compared with an hystorical control arm of recurrent ovarian cancer patients unselected for BRCA mutation or BRCAness phenotype.

SECONDARY OUTCOMES:
Response | 36 months
  -Duration of response
Progression-free survival | 36 months
  -Progression-free survival [the diagnosis of progression will be assessed by radiological criteria; CA 125 increases alone (GCIG criteria of progression) will not be considered as progression of disease without a radiological confirmation of progression].
safety profile | 36 months
  Safety profile of trabectedin in this patient population

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Scambia, Prof, Principal Investigator — Catholic University of Sacred Heart; Domenica Lorusso, Principal Investigator — National Cancer Institute, Milan
Locations (1):
- Catholic University of Sacred Heart, Rome, Rome, Italy